CLINICAL TRIAL: NCT03221283
Title: The Intervention of Group Therapy: Music in Mood Problems of Female Amphetamine Use Disorder
Brief Title: The Application of Music Therapy in Female Amphetamine Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, Min ZHAO, Vice President, Shanghai Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MZhao-007
Record Dates: First submitted 2017-07-15; First posted 2017-07-18 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Amphetamine Addiction
Keywords: Music therapy; Depression; Emotion; Motivation
MeSH Terms: conditions — Amphetamine-Related Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Participants only accept the regular scheduled in the compulsory isolated detoxification center.
- Music therapy group (Experimental): Use randomized controlled clinical trial design.The main content of music therapy is emotional experience , emotion regulation, emotional control and emotional expression. The experimental group received 13 group music sessions over a three-month period.
  Interventions: Behavioral: Music therapy group

INTERVENTIONS:
Behavioral: Music therapy group — The experimental group received 13 group music sessions over a three-month period. Different method of music therapy will be used to improve the emotion experience, emotion regulation, emotional control and emotional expression.
  Arms: Music therapy group

SUMMARY:
The group music therapy will be used to treat female amphetamine-type stimulant (ATS) addiction

DETAILED DESCRIPTION:
Amphetamine addicts are often accompanied by severe emotional problems and are difficult to control and regulate negative emotions by themselves.And the emotional problems are high risk factors of addicts relapse. Music therapy as the intervention is in order to improve amphetamine addicts' emotional status and the ability of emotion regulation. Self-rating Depression Scale(SDS), Self-rating Anxiety scale(SAS) will be used to investigate the emotion of participants. These methods will also be used to evaluate the efficacy of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* In accordance with the Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5) for methamphetamine (MA) use disorder
* Junior high school degree or above
* Normal vision and hearing
* Have emotional problem

Exclusion Criteria:

* Other substance abuse or dependence in recent a years (except nicotine)
* Mental impairment, Intelligence Quotient (IQ) < 70
* Mental disorders
* Physical disease

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Depression status assessed by Self-rating Depression Scale (SDS) at 4 months. | Baseline, 2 months,4 months, and 7months
  evaluate all participants' depression status by Self-rating Depression Scale (SDS)

SECONDARY OUTCOMES:
Anxiety status assessed by Self-rating Anxiety Scale (SAS) | Baseline, 2 months,4 months, and 7months
  evaluate all participants' anxiety status by Self-rating Anxiety Scale (SAS)
Change from Baseline Craving for ATS assessed by Visual Analog Scales (VAS) | Baseline, 2 months,4 months, and 7months
  evaluate all participants' craving for ATS by Visual Analog Scales (VAS)
Empathy ability assessed by Interpersonal Reactivity Index-C(IRI-C) | Baseline, 2 months,4 months, and 7months
  evaluate all participants' Empathy ability by Interpersonal Reactivity Index-C(IRI-C)
Motivation for treatment assessed by Stages of Change Readiness and Treatment Eagerness Scale(SOCRATES) | Baseline, 2 months,4 months, and 7months
  evaluate all participants' motivation for treatment assessed by Stages of Change Readiness and Treatment Eagerness Scale(SOCRATES)
Change from Baseline emotional status assessed by emotional STROOP paradigm | Baseline, 2 months,4 months, and 7months
  evaluate all participants' emotional status by emotional STROOP paradigm
Sleep status assessed by Pittsburgh Sleep Quality Index(PSQI) | Baseline, 2 months,4 months, and 7months
  evaluate all participants' sleep status by Pittsburgh Sleep Quality Index(PSQI)

CONTACTS AND LOCATIONS:
Overall Officials: Zhao min, PhD, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Women's Compulsory Isolation Detoxification Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No